CLINICAL TRIAL: NCT01769352
Title: Treatment of Post-surgical Cystoid Macular Edema With Topical Steroids Trial (TEMPEST-1)
Acronym: TEMPEST
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00074523
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Post-surgical Cystoid Macular Edema (PSCME)
Keywords: cystoid macular edema
MeSH Terms: conditions — Macular Edema | interventions — Ketorolac Tromethamine; Ketorolac; prednisolone acetate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PredA q1h WA + Kelac qid (Active Comparator): Prednisolone acetate (PredA) 1% ophthalmic solution every 1 hr while awake (WA) and Ketorolac (Kelac) 0.5% ophthlmic solution four times a day (qid)
  Interventions: Drug: PredA + Kelac
- PredA qid + Kelac qid (Active Comparator): Prednisolone acetate (PredA) 1% ophthalmic solution four times a day (qid) and Ketorolac (Kelac) 0.5% ophthlmic solution four times a day (qid)
  Interventions: Drug: PredA + Kelac

INTERVENTIONS:
Drug: PredA + Kelac — At week 12, patients will be determined to be resolved, improving/stabilized or treatment failures. Patients who have complete resolution of edema will begin treatment withdrawl. Improving/stabilizing patients will maintain current therapy. Treatment failure Group 2 patients will move to Group 3 to receive PredA q1h WA + Kelac qid starting at week 12. Treatment failure Group 1 patients will be exited from the trial so that alternative therapy can be given.
  Other Names: Acular, Acuvail; Pred Forte, Omnipred, Pred Mild

SUMMARY:
The purpose of this study is to compare the change in visual acuity of patients with post surgical cystoid macular edema who will be treated with two different regimens.

DETAILED DESCRIPTION:
Compare the mean change in BCVA over 12 weeks of Prednisolone Acetate 1% q1h (every hour) WA (While Awake) + Ketorolac 0.5% qid (four times a day) versus Prednisolone Acetate qid + Ketorolac qid for post surgical cystoid macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years
* Diagnosis of PSCME in study eye confirmed by FA showing leakage from retinal vessels resulting in pooling of dye in the fovea and Spectralis SD-OCT showing intraretinal fluid in or around the fovea.
* BCVA score in the study eye of 20/30 to 20/400 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters).
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from PSCME and not to any other reason.

Exclusion Criteria:

* Any patient who has other retinal diseases known to cause macular edema (choroidal neovascularization, vein occlusion, diabetic macular edema in the study eye). Patients with nonexudative Age Related Macular Degeneration (ARMD) or non-proliferative diabetic retinopathy without macular edema can be included in the study.
* Other reason for decreased visual acuity (such as amblyopia, foveal atrophy, optic atrophy).
* Pre-existing diagnosis of glaucoma in the study eye
* Inability to comply with study or follow up procedures
* Pregnancy (Women of child bearing age will be asked to take a urine pregnancy test prior to enrolling in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-Cataract Surgery CME (PredAq1h+ Kelac Qid) - Group 1: Patients who developed cystoid macular edema (CME) after cataract surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 1 hr while awake (WA) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
  PredA + Kelac: At week 12, patients will be determined to be resolved, improving/stabilized or treatment failures. Patients who have complete resolution of edema will begin treatment withdrawal. Improving/stabilizing patients will maintain current therapy. Treatment failure Group 1 patients will be exited from the trial so that alternative therapy can be given.
- Post-Cataract Surgery CME (PredA Qid + Kelac Qid) - Group 2: Patients who developed cystoid macular edema (CME) after cataract surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution four times a day (qid) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
  PredA + Kelac: At week 12, patients will be determined to be resolved, improving/stabilized or treatment failures. Patients who have complete resolution of edema will begin treatment withdrawal. Improving/stabilizing patients will maintain current therapy. Treatment failure Group 2 patients will move to Group 3 to receive PredA q1h WA + Kelac qid starting at week 12.
- Post-Other Surgery CME (PredA q1h + Kelac Qid) - Group 1: Patients who developed cystoid macular edema (CME) after other surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 1 hr while awake (WA) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
  PredA + Kelac: At week 12, patients will be determined to be resolved, improving/stabilized or treatment failures. Patients who have complete resolution of edema will begin treatment withdrawal. Improving/stabilizing patients will maintain current therapy. Treatment failure Group 1 patients will be exited from the trial so that alternative therapy can be given.
- Post-Other Surgery CME (PredA Qid + Kelac Qid) - Group 2: Patients who developed cystoid macular edema (CME) after other surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution four times a day (qid) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
  PredA + Kelac: At week 12, patients will be determined to be resolved, improving/stabilized or treatment failures. Patients who have complete resolution of edema will begin treatment withdrawal. Improving/stabilizing patients will maintain current therapy. Treatment failure Group 2 patients will move to Group 3 to receive PredA q1h WA + Kelac qid starting at week 12.
Period: Overall Study
Arm/Group | Post-Cataract Surgery CME (PredAq1h+ Kelac Qid) - Group 1 | Post-Cataract Surgery CME (PredA Qid + Kelac Qid) - Group 2 | Post-Other Surgery CME (PredA q1h + Kelac Qid) - Group 1 | Post-Other Surgery CME (PredA Qid + Kelac Qid) - Group 2
Started | 13 | 12 | 9 | 8
Completed | 13 | 12 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Post-Cataract Surgery Macular Edema- Group 1: Patients who developed cystoid macular edema (CME) after cataract surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 1 hr while awake (WA) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
- Post-Cataract Surgery Macular Edema- Group 2: Patients who developed cystoid macular edema (CME) after cataract surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 4 hr (qid) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
- Post-Other Surgery Macular Edema- Group 1: Patients who developed cystoid macular edema (CME) after other surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 1 hr while awake (WA) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
- Post-Other Surgery Macular Edema- Group 2: Patients who developed cystoid macular edema (CME) after other surgery and are started on Prednisolone acetate (PredA) 1% ophthalmic solution every 4 hr (qid) and Ketorolac (Kelac) 0.5% ophthalmic solution four times a day (qid)
- Total: Total of all reporting groups
Arm/Group | Post-Cataract Surgery Macular Edema- Group 1 | Post-Cataract Surgery Macular Edema- Group 2 | Post-Other Surgery Macular Edema- Group 1 | Post-Other Surgery Macular Edema- Group 2 | Total
Number analyzed (Participants) | 13 | 12 | 9 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (2.0) | 69.9 (2.4) | 66.2 (1.9) | 60.1 (4.8) | 67.4 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 8 | 5 | 26
  Male | 7 | 5 | 1 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 0 | 1 | 9
  White | 8 | 8 | 8 | 7 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 9 | 8 | 42
Number of Surgeries at the Time of Enrollment, mean+SEM [Mean (Standard Deviation); unit: surgeries] | 1.8 (0.2) | 1.4 (0.2) | 2.1 (0.4) | 2.1 (0.3) | 1.8 (0.1)
Best Corrected Visual Acuity at Baseline mean+SEM (Letter Score) [Mean (Full Range); unit: letters] — Best corrected visual acuity (BCVA) is a test which assesses visual acuity using an eye exam. Higher the number, better is the visual acuity and vice versa. The total score ranges from 5 to 100, with 100 representing the best visual acuity.
  letters | 55.7 [31 to 80] | 60.9 [29 to 75] | 53.4 [19 to 68] | 50.9 [20 to 73] | 55.8 [19 to 80]
CST at Baseline, mean+SEM (µm) [Mean (Standard Deviation); unit: µm] | 515.5 (33.9) | 447.6 (33.9) | 487.3 (33.3) | 489.1 (29.5) | 485.0 (16.9)
IOP at Baseline, mean+SEM (mmHg) [Mean (Standard Deviation); unit: mmHg] | 14.2 (1.3) | 15.6 (0.8) | 14.8 (0.9) | 16.0 (2.2) | 15.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best-Corrected Visual Acuity at Week 12 From Baseline
Description: Mean change in best-corrected visual acuity (Letter Score) at Week 12 from Baseline. The Early Treatment of Diabetic Retinopathy Study (ETDRS) score is measured on a scale from 5 to 100. The higher the score on this scale, the better is the patients vision.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Error); unit: letters
Arm/Group | Post-Cataract Surgery Macular Edema- Group 1 | Post-Cataract Surgery Macular Edema- Group 2 | Post-Other Surgery Macular Edema- Group 1 | Post-Other Surgery Macular Edema- Group 2
Number analyzed (Participants) | 13 | 12 | 9 | 8
letters | 10.6 (2.6) | 7.8 (3.4) | 13.1 (3.4) | 9.4 (3.6)

2. Secondary Outcome: Mean Change in Central Subfield Thickness at Week 12 From Baseline
Description: Mean Change in Central Subfield Thickness (µm) at Week 12 from Baseline
Time Frame: Baseline and Week 12
Measure: Mean (Standard Error); unit: µm
Arm/Group | Post-Cataract Surgery Macular Edema- Group 1 | Post-Cataract Surgery Macular Edema- Group 2 | Post-Other Surgery Macular Edema- Group 1 | Post-Other Surgery Macular Edema- Group 2
Number analyzed (Participants) | 13 | 12 | 8 | 8
µm | -152.7 (33.5) | -56.4 (21.0) | -25.9 (25.7) | -75.0 (30.7)

3. Secondary Outcome: Mean Change in Intraocular Pressure at Week 12 From Baseline
Description: Mean Change in Intraocular Pressure (IOP) at week 12 from Baseline
Time Frame: Baseline and Week 12
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Post-Cataract Surgery Macular Edema- Group 1 | Post-Cataract Surgery Macular Edema- Group 2 | Post-Other Surgery Macular Edema- Group 1 | Post-Other Surgery Macular Edema- Group 2
Number analyzed (Participants) | 13 | 12 | 9 | 8
mmHg | 2.6 (1.2) | 3.3 (1.4) | 0.3 (1.6) | 1.5 (1.4)

4. Secondary Outcome: Mean Change in Best-Corrected Visual Acuity Between Week 12 and Week 48
Description: Mean Change in Best-Corrected Visual Acuity (Letters Score) between Week 12 and Week 48. The Early Treatment of Diabetic Retinopathy Study (ETDRS) score is measured on a scale from 5 to 100. The higher the score on this scale, the better is the patients vision.
Time Frame: Week 12 and Week 48
Measure: Mean (Standard Error); unit: Letters
Groups:
- Prednisolone Acetate Switched From 4 Hours to Every 1 Hour: Patients who switched from Prednisolone acetate (PredA) 1% ophthalmic solution every 4 hours to every 1 hour while awake at week 12.
- Prednisolone Acetate Continued Every 1 Hour: Patients who continued on Prednisolone Acetate (PredA) 1% ophthalmic solution continued every 1 hour while awake at week 12.
- Prednisolone Acetate Switched From Every 1 Hour to 4 Hours: Patients who switched from Prednisolone Acetate (PredA) 1% ophthalmic solution from every 1 hours while awake to every 4 hours at week 12.
Arm/Group | Prednisolone Acetate Switched From 4 Hours to Every 1 Hour | Prednisolone Acetate Continued Every 1 Hour | Prednisolone Acetate Switched From Every 1 Hour to 4 Hours
Number analyzed (Participants) | 7 | 7 | 6
Letters | 9.3 (2.5) | 5.4 (2.1) | 10.8 (5.1)

5. Secondary Outcome: Mean Change in Central Subfield Thickness (CST) Between Week 12 and Week 48
Description: Mean Change in Central Subfield Thickness (CST,µm) between week 12 and week 48
Time Frame: Week 12 and Week 48
Measure: Mean (Standard Error); unit: µm
Arm/Group | Prednisolone Acetate Switched From 4 Hours to Every 1 Hour | Prednisolone Acetate Continued Every 1 Hour | Prednisolone Acetate Switched From Every 1 Hour to 4 Hours
Number analyzed (Participants) | 7 | 7 | 6
µm | -109.7 (50.9) | -44.0 (20.8) | -1.3 (6.2)

6. Secondary Outcome: Mean Change in Intraocular Pressure Between Week 12 and Week 24
Description: Mean Change in Intraocular Pressure (IOP) between week 12 and week 24
Time Frame: Week 12 and Week 48
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Prednisolone Acetate Switched From 4 Hours to Every 1 Hour | Prednisolone Acetate Continued Every 1 Hour | Prednisolone Acetate Switched From Every 1 Hour to 4 Hours
Number analyzed (Participants) | 7 | 7 | 6
mmHg | 2.3 (2.5) | 0.0 (1.7) | -4.7 (4.0)

ADVERSE EVENTS:
Time Frame: 48 Weeks
Groups:
- Prednisolone Acetate Every 1 Hour While Awake (Group 1): Patients who were given Prednisolone Acetate (PredA) 1% ophthalmic solution every 1 hour while awake.
  Adverse events are dose dependent and they don't depend on the type of surgery patient underwent previously. Therefore both, post-cataract surgery macular edema and post-other surgery macular edema adverse events were clumped together for patients who received PredA every 1 hour (q1h) - Group 1.
- Prednisolone Acetate Four Times a Day (Group 2): Patients who were given Prednisolone Acetate (PredA) 1% ophthalmic solution four times a day
  Adverse events are dose dependent and they don't depend on the type of surgery patient underwent previously. Therefore both, post-cataract surgery macular edema and post-other surgery macular edema adverse events were clumped together for patients who received PredA four times a day (qid) - Group 2.
Arm/Group | Prednisolone Acetate Every 1 Hour While Awake (Group 1) | Prednisolone Acetate Four Times a Day (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 5/22 | 4/20
Other Adverse Events (participants affected / at risk) | 6/22 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone Acetate Every 1 Hour While Awake (Group 1) (N=22) | Prednisolone Acetate Four Times a Day (Group 2) (N=20)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Blood transfusion due to severe anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Periodontal surgery (General disorders) | 1 (1) | 1 (1)
Surgery for resection of Zenker's Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cataract Surgery due to progression of cataract (Eye disorders) | 1 (1) | 1 (1)
Intraocular Pressure Lowering Surgery (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone Acetate Every 1 Hour While Awake (Group 1) (N=22) | Prednisolone Acetate Four Times a Day (Group 2) (N=20)
Increase in Intraocular Pressure (Eye disorders) | 3 (3) | 5 (5)
Upper Respiratory Tract Infections (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes